CLINICAL TRIAL: NCT01316549
Title: Population Pharmacokinetics of Fludarabine in Pediatric Patients Undergoing Hematopoietic Cell Transplantation
Brief Title: Study of Fludarabine Drug Exposure in Pediatric Bone Marrow Transplantation
Acronym: HCT
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Other Study IDs: P0037192; 10081 (Other: University of California, San Francisco)
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Hematologic Malignancies; Nonmalignant Diseases; Immunodeficiencies; Hemoglobinopathies; Genetic Inborn Errors of Metabolism; Fanconi Anemia; Thalassemia; Sickle Cell Disease
Keywords: fludarabine; pharmacokinetics; pediatric; allogeneic; hematopoietic cell transplantation
MeSH Terms: conditions — Hematologic Neoplasms; Immunologic Deficiency Syndromes; Hemoglobinopathies; Fanconi Anemia; Thalassemia; Anemia, Sickle Cell | interventions — fludarabine; fludarabine phosphate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Inpatient Pediatric Bone Marrow Transplant Recipients: All patients enrolled in this study will be located on the inpatient pediatric bone marrow transplant unit at University of California, San Francisco Benioff Children's Hospital.
  Interventions: Drug: Fludarabine

INTERVENTIONS:
Drug: Fludarabine — Given as injection
  Other Names: Fludara

SUMMARY:
Fludarabine is a chemotherapy drug used extensively in bone marrow transplantation. The goal of this study is to determine what causes some children to have different drug concentrations of fludarabine in their bodies and if drug levels are related to whether or not a child experiences severe side-effects during their bone marrow transplant. The hypothesis is that clinical and genetic factors cause changes in fludarabine drug levels in pediatric bone marrow transplant patients and that high levels may cause severe side-effects.

DETAILED DESCRIPTION:
Fludarabine is a nucleoside analog with potent antitumor and immunosuppressive properties used in conditioning regimens of pediatric allogeneic hematopoietic cell transplantation (alloHCT) to promote stem cell engraftment.

This is a single-center, pharmacokinetic-pharmacodynamic (PK-PD) study investigating the clinical pharmacology of fludarabine in 45 children undergoing alloHCT at University of California, San Francisco Benioff Children's Hospital.

Patients would receive fludarabine regardless of whether or not they decide to consent to PK sampling.

Fludarabine doses will not be adjusted based on PK data.

We will apply the combination of a D-optimality-based limited sampling strategy and population PK methodologies to determine specific factors influencing fludarabine exposure in pediatric alloHCT recipients and identify exposure-response relationships.

Subjects will undergo PK sampling of plasma (f-ara-a) and intracellular (f-ara-ATP) drug concentrations over the duration of fludarabine therapy (3 to 5 days).

To evaluate sources of variability impacting fludarabine exposure clinical data will be obtained from the patient's medical chart on each day of PK sampling.

A single blood draw for the collection of DNA and genotyping of single nucleotide polymorphisms of genes involved in fludarabine activation, transport or elimination will occur in all patients.

To assess exposure-response relationships neutrophil engraftment, treatment-related toxicity, and survival data will be collected through day 100 post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Children 0-17 years of age
* Undergoing alloHCT for the treatment of malignant or nonmalignant disorder
* Receiving fludarabine-based preparative regimen

Exclusion Criteria:

* Any child 7-17 years of age unwilling to provide assent
* Parent or guardian unwilling to provide written consent

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The target population for the proposed study includes children 0-17 years of age undergoing alloHCT for the treatment of malignant and nonmalignant disorders.
  Patients receiving fludarabine over 3 to 5 days are eligible to participate.
  All patients enrolled in this study will undergo PK sampling on the inpatient pediatric BMT unit at UCSF Benioff Children's Hospital. The proposed research will not study any patients receiving fludarabine in a clinic or any other out-patient setting.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of fludarabine for HCT in pediatric patients. | 2hours post start of infusion
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of fludarabine for HCT in pediatric patients. | 3hours post start of infusion
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of fludarabine for HCT in pediatric patients. | 6hours post start of infusion
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of fludarabine for HCT in pediatric patients. | 24hours post start of infusion

SECONDARY OUTCOMES:
Event free survival according to the AUC of fludarabine | 1month post transplant
Event free survival according to the AUC of fludarabine | 3months post transplant
Event free survival according to the AUC of fludarabine | 1 year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Janel R Long-Boyle, PharmD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ivaturi V, Dvorak CC, Chan D, Liu T, Cowan MJ, Wahlstrom J, Stricherz M, Jennissen C, Orchard PJ, Tolar J, Pai SY, Huang L, Aweeka F, Long-Boyle J. Pharmacokinetics and Model-Based Dosing to Optimize Fludarabine Therapy in Pediatric Hematopoietic Cell Transplant Recipients. Biol Blood Marrow Transplant. 2017 Oct;23(10):1701-1713. doi: 10.1016/j.bbmt.2017.06.021. Epub 2017 Jul 3. PMID 28684371